CLINICAL TRIAL: NCT04595201
Title: Clinical Follow-up of Pregnant Subjects Undergoing NIPT
Status: Recruiting | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Integrated Genetics (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCMM-RND-111
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: NIPT — Non-invasive pregnancy testing

SUMMARY:
To obtain pregnancy outcome data from patients screened for fetal genetic status using non-invasive pregnancy testing (NIPT).

DETAILED DESCRIPTION:
To obtain pregnancy outcome data from patients screened for fetal genetic status using non-invasive pregnancy testing (NIPT) to analyze the performance of routine assay enhancements and to identify characteristics associated with adverse obstetric outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subject was pregnant and received NIPT from Sequenom/Integrated Genetics
* Subject was 18 years of age or older at the time of NIPT
* Pregnancy outcome is available

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Follow-up of pregnant subjects who have undergone NIPT
Study Population: The Study Population will consist of women 18 years of age and older who underwent testing with a Sequenom NIPT and whose pregnancies should have outcome based upon gestational age at the time of testing.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2025-10-13 (Estimated)

PRIMARY OUTCOMES:
NIPT clinical outcome performance | 9 months
  Sensitivity
NIPT clinical outcome performance | 9 months
  Specificity
NIPT clinical outcome performance | 9 months
  Positive predictive value
NIPT clinical outcome performance | 9 months
  Negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Fanelli, MS, CGC, Principal Investigator — Integrated Genetics
Locations (1):
- Integrated Genetics, Westborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No